CLINICAL TRIAL: NCT02886858
Title: tDCS as Continuation Treatment to Sustain Remission After Electroconvulsive Therapy in Depression
Brief Title: tDCS in the Prevention of Relapse After Electroconvulsive Therapy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: investigator and sponsor decided by mutual agreement to stop study prematurely
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2016-A00824-47
Record Dates: First submitted 2016-08-29; First posted 2016-09-01 (Estimated); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Depression
Keywords: Depression; Moods disorders; electroconvulsive therapy
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tDCS (Experimental): The anode will be applied over the F3 area and the cathode over the F4 area. The current dose is 2mA. Electrodes will be 7x5cm in size. The investigators will apply 2 daily, tDCS sessions of 30 minutes, weekly the first month, fortnightly the second and third month, monthly the following 3 months.
  Interventions: Device: Device : Transcranial direct current stimulation
- Sham tDCS (Sham Comparator): The anode will be applied over the F3 area and the cathode over the F4 area. Electrodes will be 7x5cm in size. The investigators will apply 2 daily, tDCS sessions of 30 minutes, weekly the first month, fortnightly the second and third month, monthly the following 3 months.
  Interventions: Device: Device : sham Transcranial direct current stimulation

INTERVENTIONS:
Device: Device : Transcranial direct current stimulation — The anode will be applied over the F3 area and the cathode over the F4 area. The current dose is 2mA. Electrodes will be 7x5cm in size. The investigators will apply 2 daily, tDCS sessions of 30 minutes, weekly the first month, fortnightly the second and third month, monthly the following 3 months.
  Arms: tDCS
Device: Device : sham Transcranial direct current stimulation — The anode will be applied over the F3 area and the cathode over the F4 area. Electrodes will be 7x5cm in size. The investigators will apply 2 daily, tDCS sessions of 30 minutes, weekly the first month, fortnightly the second and third month, monthly the following 3 months.
  Arms: Sham tDCS

SUMMARY:
While electroconvulsive therapy (ECT) in major depression is effective, high relapse rates and cognitive side effects limit its long-term use. There is no consensus about optimal continuation pharmacological treatments after a ECT course.

Adjunction of tDCS to pharmacological continuation treatment after ECT may decrease relapse rates.

DETAILED DESCRIPTION:
In a prospective, randomized, double blind, controlled, long-term study, investigators assign 40 depressed patients, in remission after ECT course associated to venlafaxine, with lithium adjunction after ECT course, either to tDCS or sham tDCS. Depressive symptoms and cognition were assessed after acute ECT after six months of continuation therapy.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 ans
* Remission (MADRS <10) of a major depressive episode after acute treatment with ECT + venlafaxine
* Lithium adjunction 48h after the last ECT session
* No comorbid psychiatric disorder, excluding personality disorder or nicotine dependance.
* Capacity to consent
* Sufficient comprehension of the French language

Exclusion Criteria:

* Contra-indications to tDCS
* Neurologic conditions
* Severe medical conditions.
* Pregnancy/breast-feeding.
* Current use of benzodiazepines or antipsychotics

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-02-13 (Actual); Primary Completion 2019-04-19 (Actual); Study Completion 2019-04-19 (Actual)

PRIMARY OUTCOMES:
Relapse rate 6 months after remission, defined as the reappearance of a depressive syndrome, measured by a scoring MADRS >15. | 6 months
  MADRS will be assessed in each follow-up visit (weekly the first month, fortnightly the second and third month, monthly the following 3 months).

SECONDARY OUTCOMES:
Montreal Cognitive Assesment (MoCA) | basal and at 6 months
Scores on Clinical Global Impression (CGI) | after remission basal and at 6 months
Time to relapse | during 6 months

CONTACTS AND LOCATIONS:
Overall Officials: GALVAO FILIPE, PH, Principal Investigator — CH LE VINATIER
Locations (1):
- Centre Hospitalier Le Vinatier, Bron, Auvergne-Rhône-Alpes, France

IPD SHARING:
Plan to Share IPD: No